CLINICAL TRIAL: NCT03707652
Title: Three-Day Dosing NAD + Study
Brief Title: Open-label Study to Assess Increasing Levels of NAD+(Nicotinamide Adenine Dinucleotide)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: CL094
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-05

CONDITIONS: Increase in Blood Levels of Nicotinamide Adenine Dinucleotide (NAD+)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Cohort A (oral supplement A)-2 capsules (Experimental): Oral supplement A (2 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement A
- Cohort A (oral supplement B)-4 capsules (Experimental): Oral supplement B (4 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement B
- Cohort A (oral supplement C)-2 capsules (Experimental): Oral supplement C (2 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement C
- Cohort A (oral supplement A)-1 or 4 capsules (Experimental): Oral supplement A (1 or 4 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement A
- Cohort A (oral supplement D)-1 or 2 tablets (Experimental): Oral supplement D (1 or 2 tablets) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement D
- Cohort A (oral supplement D) or combination with supplement C (Experimental): Oral supplement D (1 or 2 tablets) or combination with oral supplement C (2 or 4 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement D; Dietary Supplement: Oral Supplement D in combination with oral supplement C
- Cohort B (oral supplement B)-4 capsules (Experimental): Oral supplement B (4 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement B
- Cohort B (oral supplement C)-2 capsules (Experimental): Oral supplement C (2 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement C
- Cohort B (oral supplement A)-2 capsules (Experimental): Oral supplement A (2 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement A
- Cohort B (oral supplement C)- 1 or 4 capsules (Experimental): Oral supplement C (1 or 4 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement C
- Cohort B (oral supplement D)-1 or 2 tablets (Experimental): Oral supplement D (1 or 2 tablets) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement D
- Cohort B(oral supplement D) or combination with supplement C (Experimental): Oral supplement D (1 or 2 tablets) or combination with oral supplement C (2 or 4 capsules) administered daily for 3 days
  Interventions: Dietary Supplement: Oral supplement D; Dietary Supplement: Oral Supplement D in combination with oral supplement C

INTERVENTIONS:
Dietary Supplement: Oral supplement A — 1, 2 or 4 capsules daily of oral supplement A for 3 days
  Other Names: Vitamin B3 derivative
  Arms: Cohort A (oral supplement A)-1 or 4 capsules; Cohort A (oral supplement A)-2 capsules; Cohort B (oral supplement A)-2 capsules
Dietary Supplement: Oral supplement B — 4 capsules daily of oral supplement B for 3 days
  Other Names: Vitamin B3 derivative
  Arms: Cohort A (oral supplement B)-4 capsules; Cohort B (oral supplement B)-4 capsules
Dietary Supplement: Oral supplement C — 1,2 or 4 capsules daily of oral supplement C for 3 days
  Other Names: Vitamin B3 derivative
  Arms: Cohort A (oral supplement C)-2 capsules; Cohort B (oral supplement C)- 1 or 4 capsules; Cohort B (oral supplement C)-2 capsules
Dietary Supplement: Oral supplement D — 1 or 2 tablets daily of oral supplement D for 3 days
  Other Names: Vitamin B3 derivative
  Arms: Cohort A (oral supplement D) or combination with supplement C; Cohort A (oral supplement D)-1 or 2 tablets; Cohort B (oral supplement D)-1 or 2 tablets; Cohort B(oral supplement D) or combination with supplement C
Dietary Supplement: Oral Supplement D in combination with oral supplement C — 1 or 2 tablets of oral supplement D in combination with 2 or 4 capsules of oral supplement C for 3 days
  Arms: Cohort A (oral supplement D) or combination with supplement C; Cohort B(oral supplement D) or combination with supplement C

SUMMARY:
The purpose of this study is to assess an effective single oral supplement or combination of oral supplements for increasing whole blood NAD+ levels.

DETAILED DESCRIPTION:
This is a open-label dose finding study to detect an effective single oral supplement or combination of oral supplements for enhancing whole blood levels of NAD+. Each subject will receive a specific dose of the formulation once daily for 3 days followed by a washout period. Upon completion of the treatment phase, there is a post-treatment period of assessments.

Participants receive assessments of blood tests, vital signs, body weight with completion of questionnaires.

The primary objective of the study is to identify the ideal dosage of an oral supplement to increase whole blood NAD+ levels in adults.

The secondary objective of the study is to monitor for safety from a change in fasting blood chemistry panel parameters after three day's dosing compared to cycle baseline.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written Informed Consent
* Able to follow verbal and written study directions in English
* Adult men and women between age 30-80 years (inclusive)
* Women of reproductive potential will practice contraception during the Investigation
* Body Mass Index (BMI) between 18.5 and 35 kg/m2
* Must not be taking or be willing to stop taking any supplements containing any form of niacin for seven days prior to baseline and for the duration of the study.
* Must not be using or be willing to stop use of any "100%" or higher niacin fortified foods from seven days prior to screening visit and for the duration of the investigation
* Able to maintain consistent diet and lifestyle habits throughout the study
* Volunteers with chronic but stable and well controlled medical conditions (i.e., hypertension controlled by a consistent dose of medication for a minimum of six months; chronic use of consistent dose of blood-thinning medication; diet-controlled Type II diabetes) may participate at the discretion of the PI or Sub-I.
* Willing and able to provide fasting blood samples
* Able to attend scheduled visits at the Life Extension Clinical Research (LECR) facility

Exclusion Criteria:

* Current use of prescription or over-the-counter nicotinic acid
* Use of statin drugs
* Having used any tobacco product or used a recreational drug in the past 6 months
* Medically complicated [i.e., diabetes requiring insulin; uncontrolled hypertension (blood pressure readings at screening/baseline > 140 systolic or > 90 diastolic on two consecutive readings); etc.] at the discretion of the PI or Sub-I
* Having abnormal screening laboratory test values or other lab test result(s) that would preclude study participation in the judgment of the PI or Sub-I
* Woman who is pregnant, nursing, or planning a pregnancy. Non-pregnant status of women of childbearing potential will be confirmed during each Day 3 Cycle LECR visit (Wednesday or Thursday) via serum pregnancy test.
* Currently, or within the past 30 days, enrolled in a different clinical investigation
* Inability to provide a venous blood sample
* Unable to refrain from any alcohol consumption for the duration of the study
* Unable or unwilling to provide written informed consent for participation in study

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Assess the mean change in NAD+ levels from baseline | 63 days
  Mean change in NAD+ levels

SECONDARY OUTCOMES:
Assess the mean change in AST (aspartate aminotransferase) levels from baseline | 63 days
  Mean change in AST level
Assess the mean change in ALT (alanine aminotransferase) levels from baseline | 63 days
  Mean change in ALT level
Assess the mean change in Total Cholesterol levels from baseline | 63 days
  Mean change in Total Cholesterol level
Assess the mean change in Triglycerides levels from baseline | 63 days
  Mean change in Triglycerides level
Assess the mean change in LDL Cholesterol levels from baseline | 63 days
  Mean change in LDL Cholesterol level
Assess the mean change in HDL Cholesterol levels from baseline | 63 days
  Mean change in HDL Cholesterol level

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, Ph.D, Principal Investigator — LIfe Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kennedy BK, Berger SL, Brunet A, Campisi J, Cuervo AM, Epel ES, Franceschi C, Lithgow GJ, Morimoto RI, Pessin JE, Rando TA, Richardson A, Schadt EE, Wyss-Coray T, Sierra F. Geroscience: linking aging to chronic disease. Cell. 2014 Nov 6;159(4):709-13. doi: 10.1016/j.cell.2014.10.039. PMID 25417146
- [Background] Massudi H, Grant R, Braidy N, Guest J, Farnsworth B, Guillemin GJ. Age-associated changes in oxidative stress and NAD+ metabolism in human tissue. PLoS One. 2012;7(7):e42357. doi: 10.1371/journal.pone.0042357. Epub 2012 Jul 27. PMID 22848760
- [Background] Verdin E. NAD(+) in aging, metabolism, and neurodegeneration. Science. 2015 Dec 4;350(6265):1208-13. doi: 10.1126/science.aac4854. PMID 26785480
- [Background] Revollo JR, Grimm AA, Imai S. The regulation of nicotinamide adenine dinucleotide biosynthesis by Nampt/PBEF/visfatin in mammals. Curr Opin Gastroenterol. 2007 Mar;23(2):164-70. doi: 10.1097/MOG.0b013e32801b3c8f. PMID 17268245
- [Background] Yang H, Lavu S, Sinclair DA. Nampt/PBEF/Visfatin: a regulator of mammalian health and longevity? Exp Gerontol. 2006 Aug;41(8):718-26. doi: 10.1016/j.exger.2006.06.003. Epub 2006 Jul 13. PMID 16842957
- [Background] Gross CJ, Henderson LM. Digestion and absorption of NAD by the small intestine of the rat. J Nutr. 1983 Feb;113(2):412-20. doi: 10.1093/jn/113.2.412. PMID 6218262
- [Background] Knip M, Douek IF, Moore WP, Gillmor HA, McLean AE, Bingley PJ, Gale EA; European Nicotinamide Diabetes Intervention Trial Group. Safety of high-dose nicotinamide: a review. Diabetologia. 2000 Nov;43(11):1337-45. doi: 10.1007/s001250051536. PMID 11126400
- [Background] Airhart SE, Shireman LM, Risler LJ, Anderson GD, Nagana Gowda GA, Raftery D, Tian R, Shen DD, O'Brien KD. An open-label, non-randomized study of the pharmacokinetics of the nutritional supplement nicotinamide riboside (NR) and its effects on blood NAD+ levels in healthy volunteers. PLoS One. 2017 Dec 6;12(12):e0186459. doi: 10.1371/journal.pone.0186459. eCollection 2017. PMID 29211728
- [Background] Dellinger RW, Santos SR, Morris M, Evans M, Alminana D, Guarente L, Marcotulli E. Repeat dose NRPT (nicotinamide riboside and pterostilbene) increases NAD+ levels in humans safely and sustainably: a randomized, double-blind, placebo-controlled study. NPJ Aging Mech Dis. 2017 Nov 24;3:17. doi: 10.1038/s41514-017-0016-9. eCollection 2017. PMID 29184669
- [Background] Trammell SA, Schmidt MS, Weidemann BJ, Redpath P, Jaksch F, Dellinger RW, Li Z, Abel ED, Migaud ME, Brenner C. Nicotinamide riboside is uniquely and orally bioavailable in mice and humans. Nat Commun. 2016 Oct 10;7:12948. doi: 10.1038/ncomms12948. PMID 27721479
- [Background] de Picciotto NE, Gano LB, Johnson LC, Martens CR, Sindler AL, Mills KF, Imai S, Seals DR. Nicotinamide mononucleotide supplementation reverses vascular dysfunction and oxidative stress with aging in mice. Aging Cell. 2016 Jun;15(3):522-30. doi: 10.1111/acel.12461. Epub 2016 Mar 11. PMID 26970090
- [Background] Mills KF, Yoshida S, Stein LR, Grozio A, Kubota S, Sasaki Y, Redpath P, Migaud ME, Apte RS, Uchida K, Yoshino J, Imai SI. Long-Term Administration of Nicotinamide Mononucleotide Mitigates Age-Associated Physiological Decline in Mice. Cell Metab. 2016 Dec 13;24(6):795-806. doi: 10.1016/j.cmet.2016.09.013. Epub 2016 Oct 27. PMID 28068222
- [Background] ClinicalTrials.gov. Effect of
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes and its Panel on Folate, Other B Vitamins, and Choline. Dietary Reference Intakes for Thiamin, Riboflavin, Niacin, Vitamin B6, Folate, Vitamin B12, Pantothenic Acid, Biotin, and Choline. Washington (DC): National Academies Press (US); 1998. Available from http://www.ncbi.nlm.nih.gov/books/NBK114310/ PMID 23193625